CLINICAL TRIAL: NCT00560222
Title: Randomized, Controlled Trial - Lactoferrin Prevention of Diarrhea in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Thomas G Cleary, Professor, Division of Epidemiology, Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1R01HD051716-01A2 (NIH); 1R01HD051716-01A2 (NIH)
Record Dates: First submitted 2007-11-15; First posted 2007-11-19 (Estimated); Last update posted 2011-11-01 (Estimated); Status verified 2011-10

CONDITIONS: Diarrhea; Malnutrition
Keywords: randomized controlled trial; lactoferrin; children; diarrhea; malnutrition; growth
MeSH Terms: conditions — Diarrhea; Malnutrition | interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): This group will receive daily lactoferrin supplementation
  Interventions: Dietary Supplement: bovine lactoferrin
- B (Placebo Comparator): placebo
  Interventions: Dietary Supplement: placebo [maltodextrin]

INTERVENTIONS:
Dietary Supplement: bovine lactoferrin — 1gm of lactoferrin will be given each day
  Arms: A
Dietary Supplement: placebo [maltodextrin] — placebo that appears identical to lactoferrin will be given daily
  Arms: B

SUMMARY:
Much has been learned in recent years about the mechanisms by which breastfeeding improves child health and survival. However, there has been little progress in using these insights to improve pediatric care. Factors that are important for protecting the breast fed infant might be expected to decrease the adverse effects of weaning on diarrhea, growth, and development. The proposed study is meant to begin addressing this important gap by a clinical trial of lactoferrin supplementation in previously weaned children. Lactoferrin,an iron-binding protein with multiple physiological functions (anti-microbial, anti-inflammatory, and immunomodulatory), is one of the most important proteins present in mammalian milk. Our hypothesis is that lactoferrin (given as a daily supplement in amounts similar to those consumed if the child were still breastfed) will improve health by mimicking its protective roles in milk. The significance of these studies is that they will prove feasibility of improving child health after the end of breastfeeding by continuing ingestion of a major protective milk protein. Diarrhea and malnutrition after weaning is a global problem that may be amenable to this approach.

DETAILED DESCRIPTION:
The proposed community-based study will be conducted in a previously weaned population at risk for repeated intestinal infections. Infants who are 12-18 months of age living in the District of Independencia, Lima, Peru will be eligible for enrollment. We will conduct a randomized double blind placebo controlled trial comparing twice daily supplementation with bovine lactoferrin versus a placebo (maltodextrin) Therapy will be continued for 6 months with close monitoring of all study participants for diarrhea and growth.

Specific aim 1: Determine the effect of bovine lactoferrin supplementation on prevention of diarrhea,measured by the number of episodes of diarrhea during a 6 month trial in previously weaned Peruvian children enrolled at 12 to 18 months of age.

Specific aim 2: Determine the effect of bovine lactoferrin supplementation on growth.

ELIGIBILITY:
Inclusion Criteria:

1. Infants 12 to 18 months of age from the Outpatient clinics (Puestos de Salud) of Districto de Independencia in Lima, Peru will be eligible for enrollment in this study.
2. Infants previously weaned for at least one week will be eligible for study.

Exclusion Criteria:

1. Infants with either exclusive or partial breast-feeding will not be enrolled; mothers will be encouraged to continue breastfeeding.
2. Infants ill with severe, persistent or chronic diarrhea will be excluded.
3. Infants with severe malnutrition (defined as weight-for-height < -3 SDs, height-for-age < -3SDs)will be excluded.
4. Infants with a serious infections that required hospitalization 1 month prior (e.g. meningitis,pneumonia, bacteremia) will be excluded.
5. Infants with known HIV (data from parent or medical records) will be excluded.
6. Infants with underlying chronic illness (e.g. malignancy, immunosuppression, chronic renal failure, congestive heart failure, liver failure) will be excluded.
7. Infants with history of allergy to cow's milk or infant formula, eczema, allergic rhinitis or asthma will be excluded.
8. Infants with a family history of eczema, allergic rhinitis, asthma, or milk intolerance will be excluded.

Ages: 12 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 555 (Actual)
Dates: Start 2008-02; Primary Completion 2011-05 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Determination of the effect of bovine lactoferrin supplementation on prevention of diarrhea,measured by the number of episodes of diarrhea during a 6 month trial in previously weaned Peruvian children enrolled at 12 to 18 months of age. | 6 months

SECONDARY OUTCOMES:
Determination of the effect of bovine lactoferrin supplementation on growth. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas G Cleary, MD, Principal Investigator — University of Texas School of Public Health - Houston
Locations (1):
- Universidad Peruana Cayetana Heredia, Lima, Peru

REFERENCES:
- [Background] Ochoa TJ, Noguera-Obenza M, Cleary TG. Lactoferrin blocks the initial host cell attachment mechanism of Enteropathogenic E. coli (EPEC). Adv Exp Med Biol. 2004;554:463-6. doi: 10.1007/978-1-4757-4242-8_65. No abstract available. PMID 15384625
- [Background] Ochoa TJ, Noguera-Obenza M, Ebel F, Guzman CA, Gomez HF, Cleary TG. Lactoferrin impairs type III secretory system function in enteropathogenic Escherichia coli. Infect Immun. 2003 Sep;71(9):5149-55. doi: 10.1128/IAI.71.9.5149-5155.2003. PMID 12933858
- [Background] Ochoa TJ, Brown EL, Guion CE, Chen JZ, McMahon RJ, Cleary TG. Effect of lactoferrin on enteroaggregative E. coli (EAEC). Biochem Cell Biol. 2006 Jun;84(3):369-76. doi: 10.1139/o06-053. PMID 16936809
- [Background] Gomez HF, Ochoa TJ, Carlin LG, Cleary TG. Human lactoferrin impairs virulence of Shigella flexneri. J Infect Dis. 2003 Jan 1;187(1):87-95. doi: 10.1086/345875. Epub 2002 Dec 13. PMID 12508150
- [Background] Gomez HF, Ochoa TJ, Herrera-Insua I, Carlin LG, Cleary TG. Lactoferrin protects rabbits from Shigella flexneri-induced inflammatory enteritis. Infect Immun. 2002 Dec;70(12):7050-3. doi: 10.1128/IAI.70.12.7050-7053.2002. PMID 12438385
- [Background] Gomez HF, Herrera-Insua I, Siddiqui MM, Diaz-Gonzalez VA, Caceres E, Newburg DS, Cleary TG. Protective role of human lactoferrin against invasion of Shigella flexneri M90T. Adv Exp Med Biol. 2001;501:457-67. doi: 10.1007/978-1-4615-1371-1_57. PMID 11787716
- [Derived] Ochoa TJ, Chea-Woo E, Baiocchi N, Pecho I, Campos M, Prada A, Valdiviezo G, Lluque A, Lai D, Cleary TG. Randomized double-blind controlled trial of bovine lactoferrin for prevention of diarrhea in children. J Pediatr. 2013 Feb;162(2):349-56. doi: 10.1016/j.jpeds.2012.07.043. Epub 2012 Aug 30. PMID 22939927